CLINICAL TRIAL: NCT07162701
Title: Body Composition Assessment and Monitoring With Bioelectrical Impedance Analysis to Predict Medical Therapy Efficacy in Inflammatory Bowel Disease (the BAMBIE Study)
Brief Title: Body Composition Assessment and Monitoring in Inflammatory Bowel Disease
Acronym: BAMBIE
Status: Recruiting | Type: Observational
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Grupo Español de trabajo en Enfermedad de Crohn y Colitis Ulcerosa (GETECCU) (Unknown)
Responsible Party: Sponsor
Other Study IDs: IIBSP-DAM-2024-216
Record Dates: First submitted 2025-08-06; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Body Composition Changes; Malnutrition
Keywords: malnutrition; IBD; BIA; composition; body; Crohn; colitis
MeSH Terms: conditions — Malnutrition; Colitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ulcerative colitis: Pacients with ulcerative colitis
  Interventions: Diagnostic Test: Bioimpedance analysis
- Crohn's disease: Patients with Crohn's disease
  Interventions: Diagnostic Test: Bioimpedance analysis

INTERVENTIONS:
Diagnostic Test: Bioimpedance analysis — Patients' body composition will be assessed using bioimpedance analysis (Akern)

SUMMARY:
This is a single-center, prospective observational study aiming to describe changes in body composition (specifically, percentage of lean mass and phase angle) in patients with active inflammatory bowel disease (IBD), including ulcerative colitis and Crohn's disease.

The study will recruit patients with a confirmed IBD diagnosis who are starting biologic therapy or Janus kinase inhibitors (JAKi) to induce clinical remission. Body composition will be assessed using bioelectrical impedance analysis (BIA) at baseline (time 0), 24 weeks, and 52 weeks after starting medication. Clinical disease activity, endoscopic findings, and laboratory data will also be collected at various time points if available.

The study has a total duration of 36 months, including a 12-18 month patient inclusion period and a 12-month follow-up. Patients will provide informed consent, and all treatment decisions will follow standard clinical practice, as this is a non-interventional observational study.

ELIGIBILITY:
Inclusion Criteria:

* Any sex.
* Age between 18 and 64 years.
* Patients with a definitive diagnosis (>3 months) of Crohn's disease or ulcerative colitis, according to European Crohn's and Colitis Organization criteria.
* Moderate-to-severe disease luminal activity, with an indication for biologic or JAKi therapy for the induction of clinical remission.

Exclusion Criteria:

* Unclassified IBD.
* History of intestinal resection for IBD, with the exception of ileocecal resection.
* Short bowel syndrome.
* Indication for medical treatment due to postsurgical recurrence.
* Active perianal disease.
* Indication for medical treatment due to intestinal stricture.
* Previous participation in a clinical trial involving medication for IBD treatment.
* Engaging in vigorous physical activity (>6 Metabolic Equivalent of Task, METs) for more than 3 days per week.
* Habitual alcohol consumption (>1 standard drink unit/day).
* Diabetes mellitus with inadequate glycemic control.
* Chronic use of diuretics.
* Chronic kidney disease on dialysis.
* Presence of dependent edema and/or ascites.
* Cardiac pacemaker bearers.
* Pregnant or lactating women.
* Inability to sign informed consent.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with IBD (Crohn's disease and ulcerative colitis)
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2026-07-15 (Estimated); Study Completion 2028-07-15 (Estimated)

PRIMARY OUTCOMES:
Phase angle change | 24 weeks
  To describe the changes in Phase angle observed between week 0 (baseline) and week 24 after the commencement of biologic or JAK inhibitor therapy.
Body Composition change | 24 months
  To describe the changes in Lean Mass index observed between week 0 (baseline) and week 24 after the commencement of biologic or JAK inhibitor therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Unidad de Enfermedad Inflamatoria Intestinal, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
Due to local privacy regulations, data can only be shared upon written, motivated request and approval by the local IEC.